CLINICAL TRIAL: NCT01415492
Title: Multiple Risk Behavior Intervention in Health Care Settings
Acronym: HD2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Emmons, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1810; 5R01CA123228 (NIH)
Record Dates: First submitted 2011-08-10; First posted 2011-08-12 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Health Behavior; Risk Reduction Behavior
Keywords: Exercise; Physical activity; Cigarette Smoking; Smoking cessation; Multi Vitamin intake; Vegetable consumption; Fruit consumption; Meat consumption
MeSH Terms: conditions — Health Behavior; Risk Reduction Behavior; Motor Activity; Cigarette Smoking; Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): At recruitment this group only received five pamphlets from the study. Four of these pamphlets were from the American Cancer Society, and one from Quitworks (a smoking cessation program).
- HD2 (Active Comparator): The intervention study information was delivered via print materials or access to a HD2 Web Site. Patients chose modality. ADDITIONAL NOTE: A sub-set of these participants was randomly selected to receive the Electronic Reminders through the intervention.
  Interventions: Behavioral: HD2
- HD2+ (Active Comparator): The intervention study information was delivered via print materials or access to a HD2 Web Site. Patients chose modality. In addition participants received two coaching calls from Health Coaches. ADDITIONAL NOTE: A sub-set of these participants was randomly selected to receive the Electronic Reminders through the intervention.
  Interventions: Behavioral: HD2+

INTERVENTIONS:
Behavioral: HD2 — The intervention was delivered via either print materials or access to a HD2 Web Site. ADDITIONAL NOTE: A sub-set of these participants was randomly selected to receive the Electronic Reminders through the intervention. Those who were selected could choose to receive the Electronic Reminders either as text messages or as automated phone reminders.
  Arms: HD2
Behavioral: HD2+ — The intervention was delivered via either print materials or access to a HD2 Web Site. In addition participants received two coaching calls from Health Coaches. ADDITIONAL NOTE: as noted above, a sub-set of these participants was randomly selected to receive the Electronic Reminders through the intervention. Those who were selected could choose to receive the Electronic Reminders either as text messages or as automated phone reminders.
  Arms: HD2+

SUMMARY:
This study (aka Healthy Directions2 or HD2) builds on an earlier study titled Healthy Directions (aka Healthy Directions 1 or HD1). HD1 was an intervention designed to target cancer prevention among multi-ethnic populations; it led to significant improvements in the multiple risk behavior score (consumption of red meat, fruits and vegetables, and multi-vitamins). Building on the success of HD1, HD2 further expanded the intervention to include smoking and physical activity. In addition, it expanded the study goals to include increasing efficacy across all target risk behaviors, and promoting long-term maintenance of behavior change.

DETAILED DESCRIPTION:
HD2 conducted a randomized control trial at two metropolitan Harvard Vanguard Medical Associates (HVMA) sites. The unit of randomization was the primary care provider. Providers were randomized to one of three arms:

1. Usual care, a control arm.
2. HD2, an intervention arm, which included access to the study information via website or study information content via print materials. Content addressed the 5 targeted health behaviors and goals, the importance of tracking behaviors in order to improve behaviors, and the importance of social support during behavior change.
3. HD2+, another intervention arm, which included access to the study information content just described, PLUS two coaching calls.

Note: access to the website was available for the 6 months after recruitment only.

In addition, the investigators wanted to test how use of electronic reminders might increase engagement with the intervention. So, a sub-set of both intervention arms was randomized to receive additional electronic reminders. Participants were allowed to choose either AVR (voicemail) or SMS (text messaging) for the delivery of these brief electronic reminders.

The investigators conducted recruitment on a rolling basis. Patients were assigned to the conditions to which their primary care providers were randomized. The investigators offered participation to providers from the Internal Medicine departments who had full patient panels and conducted annual well visit physicals with adult HVMA patients. All participating providers were informed about the HD2 study through a presentation by study staff. Providers could elect to opt out of participation prior to the patient recruitment period.

Potentially eligible patients were sent a recruitment letter before their appointment date. This letter introduced the study and let patients know that study staff may approach them at the clinic to further discuss possible participation. The letter also included a phone number for patients to call if they wanted to opt-out of being approached.

At the appointment, study staff approached people who did not opt out. They discussed the study, answered any questions, screened for eligibility, and then enrolled interested, eligible patients. Once patients signed the informed consent they were asked to complete a written, self-administered, baseline survey and given a small incentive for their time.

After completing the baseline survey, patients in the UC group only received 5 pamphlets addressing the 5 behaviors of the study. In addition to the study materials described previously, HD2 and HD2+ participants received a bottle of multi-vitamins and pedometer to support these two health behaviors. HD2 and HD2+ participants also received a tailored feedback report based on their baseline survey responses (mailed to participants approximately one week post recruitment).

All participants who completed the baseline survey were contacted for two follow-up surveys, which were administered over the phone by survey assistants. The first follow-up survey was done at the end of their intervention period (6 months post recruitment). The second follow-up survey was done at 18 months post recruitment). Those participants who were unreachable by telephone were given the option to complete an abbreviated version of the survey, which was sent to them via the mail. A small incentive was given to participants after completion of each follow-up survey.

AIMS:

A.1. To determine the efficacy of the HD2 intervention. Hypothesis 1.1: Participants in HD2/HD2+ interventions will achieve significantly greater change in the multiple risk behavior score at 6- and 18-month follow-ups than those UC.

Hypothesis 1.2: Participants in HD2/HD2+ interventions will achieve significantly greater change in individual risk factors at 6- and 18-month follow-ups, compared to those in UC (secondary outcomes).

Hypothesis 1.3: Participants who receive electronic reminders will achieve significantly greater change in the multiple risk behavior score at 6- and 18-month follow-ups than those who do not.

Hypothesis 1.4: Participants who receive electronic reminders will achieve significantly greater change in individual risk factors at 6- and 18-month follow-ups than those who do not.

A.2. To evaluate the impact of the HD2/HD2+ intervention in terms of maximizing participation/reach, intervention delivery, and cost-effectiveness.

A3. To determine whether providing assistance with a key component of the web site, behavior tracking, will stimulate higher rates of use.

Validation component of the parent study: N = 150 participants. As part of the protocol, the investigators recruited a small sample from the original cohort. All quit smokers were offered enrollment and a random sample of the remaining cohort was offered enrollment. The investigators used "gold standards" to validate these data. Dietary data (fruit & vegetable, red meat, multivitamin use) were measured by 24-hour telephone-administered food recall interviews. Physical activity was measured by accelerometers. Smoking cessation was measured by saliva cotinine testing.

TRACKING SUBSTUDY (n=100)

Aim of substudy:

To determine whether providing assistance with a key component of the web site, behavior tracking, will stimulate higher rates of use.

Methods:

All eligible and interested participants will be enrolled recruited into the web arm of the parent study intervention only. We will use the same eligibility criteria and data collection.

In summary, self-monitoring rates of enrolled patients will be assessed at day 7 for HD2 website use. If he/she has logged into the HD2 web site and completed behavior tracking at least 3 times they will continue in the study with no additional technical support. Participants who have not completed behavior self-monitoring at least 3 times will then be divided into two groups. Group 1 will receive Automated Assistance (emails) only and Group 2 will receive Personal Assistance (2 calls from trained staff offering technical assistance if needed) & Automated Assistance emails like Group 1.

ELIGIBILITY:
Inclusion Criteria:

* HVMA patient seeing a provider participating in HD2 for annual well visit
* 18 years of age or older
* Able to read in English

Exclusion Criteria:

* No diagnosis of dementia or psychotic disorders
* Undergone cancer treatment within past year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2440 (Actual)
Dates: Start 2009-03; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in multiple risk behavior (MRB) score | 6- and 18- months post intervention follow-ups
  Change in multiple risk behavior (MRB) score at the 6- and 18-months post-intervention follow-ups. This score is a composite measure comprised of status on 5 individual risk factors: red meat intake, multi-vitamin intake, and fruit and vegetable intake, physical activity, and smoking cessation

SECONDARY OUTCOMES:
Change in each of the target risk factors | 6- and 18- months post intervention follow-ups
  Change in each of the target risk factors intervention dose delivered, reach, and cost-effectiveness.

OTHER OUTCOMES:
Tracking substudy | starting 7 days after enrollment into the study
  To determine whether providing assistance with a key component of the web site, behavior tracking, will stimulate higher rates of use.

CONTACTS AND LOCATIONS:
Overall Officials: Karen M. Emmons, Ph.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Harvard Vanguard Medical Associates, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Greaney ML, Puleo E, Bennett GG, Haines J, Viswanath K, Gillman MW, Sprunck-Harrild K, Coeling M, Rusinak D, Emmons KM. Factors associated with choice of web or print intervention materials in the healthy directions 2 study. Health Educ Behav. 2014 Feb;41(1):52-62. doi: 10.1177/1090198113486803. Epub 2013 May 29. PMID 23720532
- [Background] Lewis KH, Gillman MW, Greaney ML, Puleo E, Bennett GG, Emmons KM. Relationships between Social Resources and Healthful Behaviors across the Age Spectrum. J Aging Res. 2012;2012:501072. doi: 10.1155/2012/501072. Epub 2012 Aug 30. PMID 22970369
- [Result] Greaney ML, Puleo E, Sprunck-Harrild K, Bennett GG, Cunningham MA, Gillman MW, Coeling M, Emmons KM. Electronic reminders for cancer prevention: factors associated with preference for automated voice reminders or text messages. Prev Med. 2012 Aug;55(2):151-4. doi: 10.1016/j.ypmed.2012.05.014. Epub 2012 May 30. PMID 22659227
- [Result] Greaney ML, Sprunck-Harrild K, Bennett GG, Puleo E, Haines J, Viswanath KV, Emmons KM. Use of email and telephone prompts to increase self-monitoring in a Web-based intervention: randomized controlled trial. J Med Internet Res. 2012 Jul 27;14(4):e96. doi: 10.2196/jmir.1981. PMID 22842775
- [Result] Emmons KM, Puleo E, Greaney ML, Gillman MW, Bennett GG, Haines J, Sprunck-Harrild K, Viswanath K. A randomized comparative effectiveness study of Healthy Directions 2--a multiple risk behavior intervention for primary care. Prev Med. 2014 Jul;64:96-102. doi: 10.1016/j.ypmed.2014.03.011. Epub 2014 Mar 16. PMID 24642140